CLINICAL TRIAL: NCT00088595
Title: An Open-label, Multicenter, Phase II Study Evaluating the Safety and Efficacy of Twice Daily Dosing of SOM230 in Patients With Metastatic Carcinoid Tumors
Brief Title: Study Evaluating SOM230 in Patients With Metastatic Carcinoid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230B2202
Record Dates: First submitted 2004-07-30; First posted 2004-08-02 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Carcinoid Tumors
Keywords: SOM230; Sandostatin; Carcinoid syndrome
MeSH Terms: conditions — Carcinoid Tumor; Serotonin Syndrome | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pasireotide (Experimental)
  Interventions: Drug: Pasireotide (SOM230)

INTERVENTIONS:
Drug: Pasireotide (SOM230) — Open label. Patients received starting dose of 300 µg of study drug subcutaneously (s.c.) twice (total of 600 µg ) daily for three days, which could be increased in 150 µg increments up to 900 µg twice daily (total 1800 µg daily) if control of symptoms was not achieved. Prior sponsor agreement was required for a higher dose. A dose of 2400 µg/day was the maximum allowed. Dose reductions of 300 µg/day were allowed at any time if unacceptable toxicity occurred.
  Other Names: SOM230

SUMMARY:
Study evaluating SOM230 in patients with metastatic carcinoid tumors

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven metastatic carcinoid tumors
* Patients with at least one measurable lesion (excluding bone)
* Patients must be considered inadequately controlled while on Sandostatin LAR therapy based on the symptoms of carcinoid syndrome (diarrhea and/or flushing) as defined as experiencing a minimum average of at least four bowel movements per day or a minimum average of at least two episodes of flushing per day

Exclusion Criteria:

* Patients who have been previously treated with certain medications may be required to be without certain medications prior to entering the study
* Patients who have undergone major recent surgery / surgical therapy for any cause within 1 month
* Patients on any cytotoxic chemotherapy or interferon therapy within the last 2 months
* Patients with uncontrolled diabetes mellitus
* Patients who had received radiotherapy for any reason within the last 4 weeks must have recovered from any side effects of radiotherapy
* Patients who have congestive heart failure unstable angina, cardiac arrhythmia or a history of acute myocardial infarction within the three months preceding enrollment
* Patients with chronic liver disease
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method for birth control.
* History of immunocompromise, including a positive HIV test result
* Patients who have a history of alcohol or drug abuse in the 6 month period prior to receiving SOM230
* Patients who have given a blood donation (of 400 mL or more) within 2 months before receiving SOM230
* Patients who have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Patients with additional active malignant disease within the last five years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Univ. Of Iowa Holden Cancer Center, Iowa City, Iowa
  - Louisiana State University Medical Center, New Orleans, Louisiana

RESULTS

PARTICIPANT FLOW:
Groups:
- Pasireotide (Any Dose): SOM230 (Pasireotide), 150µg twice daily dose titration up to 1200µg twice daily, subcutaneous injection.
Period: Overall Study
Arm/Group | Pasireotide (Any Dose)
Started | 45
Completed | 17
Not Completed | 28
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 8
Not completed — Ongoing (After Core) | 7
Not completed — New Cancer Therapy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pasireotide (Any Dose)
Number analyzed (Participants) | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 61.0 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 24
  Sweden | 5
  Germany | 11
  Netherlands | 4
  France | 1

OUTCOME MEASURES:

1. Primary Outcome: Symptom Control (Diarrhea/Flushing) Using a Patient Symptom Diary
Description: Complete Symptom Control: an average of ≤ 3 bowel movements per day for at least 15 consecutive days, with no more than 3 episodes on any given day, and no episodes of flushing over the time interval being studied.
  Partial Symptom Control: an average of < 4 bowel movements per day for at least 15 consecutive days, with no more than 6 episodes per given day, and an average of fewer than 2 daily flushing episodes over the same given time interval.
  Treatment failure: Failure to obtain partial or complete treatment success over a consecutive 15-day period at a constant dose level.
Time Frame: 15 days
Population: The efficacy analysis population (EAP) consisted of 44 patients all of whom had at least one efficacy assessment available after receiving at least one dose of study drug, but excluded 1 patient who had no post-baseline efficacy assessments.
Measure: Number; unit: participants
Arm/Group | Pasireotide (Any Dose)
Number analyzed (Participants) | 44
participants
  Complete symptom control | 3
  Partial symptom control | 9
  No control | 32

2. Secondary Outcome: Duration of Complete Symptom Control (Days) by Dose Class
Description: Complete symptom control: an average of three or less bowel movements per day for at least 15 consecutive days, with no more than three episodes on any given day, and no episodes of flushing over the time interval being studied.
Time Frame: 15 days
Population: The efficacy analysis population (EAP) consisted of 44 patients all of whom had at least one efficacy assessment available after receiving at least one dose of study drug, but excluded 1 patient who had no post-baseline efficacy assessments. n= the number of patients with complete symptom control.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Pasireotide 300 - ≤900 μg: SOM230 (Pasireotide), 300 - ≤900 μg / day
- Pasireotide >900 - ≤1500 μg: SOM230 (Pasireotide), >900 - ≤1500 μg / day
- Pasireotide >1500 - ≤2400 μg: SOM230 (Pasireotide), >1500 - ≤2400 μg / day
- Pasireotide Any Dose: SOM230 (Pasireotide), 300 ug - 2400 ug / day
Arm/Group | Pasireotide 300 - ≤900 μg | Pasireotide >900 - ≤1500 μg | Pasireotide >1500 - ≤2400 μg | Pasireotide Any Dose
Number analyzed (Participants) | 0 | 2 | 1 | 3
Days |  | 42.0 (22.68) | 47.0 (NA) — Upper limit not attained since there is only one observation | 43.7 (16.26)

3. Secondary Outcome: Duration of Partial Symptom Control (Days) by Dose Class
Description: Partial symptom control: an average of less than four bowel movements per day for at least 15 consecutive days, with no more than six episodes per any given day, and an average of less than two daily flushing episodes over the same given time interval.
Time Frame: up to 15 days
Population: The efficacy analysis population (EAP) consisted of 44 patients all of whom had at least one efficacy assessment available after receiving at least one dose of study drug, but excluded 1 patient who had no post-baseline efficacy assessments. n= then number of patients with partial sympton control
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Pasireotide 300-≤900 μg: SOM230 (Pasireotide), 150µg twice daily dose titration up to 450µg twice daily, subcutaneous injection.
- Pasireotide >900-≤1500 μg: SOM230 (Pasireotide), more than 450µg twice daily dose titration up to 750µg twice daily, subcutaneous injection.
- Pasireotide >1500-≤2400 μg: SOM230 (Pasireotide), more than 750µg twice daily dose titration up to 1200µg twice daily, subcutaneous injection.
- Pasireotide Any Dose: SOM230 (Pasireotide), 150µg twice daily dose titration up to 1200µg twice daily, subcutaneous injection.
Arm/Group | Pasireotide 300-≤900 μg | Pasireotide >900-≤1500 μg | Pasireotide >1500-≤2400 μg | Pasireotide Any Dose
Number analyzed (Participants) | 0 | 6 | 3 | 9
Days |  | 89.8 (95.77) | 36.3 (28.73) | 72.0 (81.58)

4. Secondary Outcome: The Number of Patients (Participants) With Overall Tumor Response
Description: The disappearance of all lesions was considered a complete response and at least a 30% decrease in the diameter of lesions was considered a partial response (PR). Progressive disease (PD) required a 20% increase in the sum of the diameters of lesions and changes that did not qualify for PR or PD were considered stable disease. Progression not documented was defined as unknown. No more than a 10% increase in biochemical values, and no clinical signs of DP with complete or adequate control over symptoms were defined as complete treatment success and partial treatment success, respectively.
Time Frame: At least 15 days
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pasireotide (Any Dose)
Number analyzed (Participants) | 44
Participants
  Complete response for complete treatment success | 0
  Partial response for complete treatment success | 0
  Stable disease for complete treatment success | 1
  Progressive disease for complete treatment success | 0
  Unknown for complete treatment success | 0
  Missing for complete treatment success | 0
  Complete response for partial treatment success | 0
  Partial response for partial treatment success | 0
  Stable disease for partial treatment success | 4
  Progressive disease for partial treatment success | 0
  Unknown for partial treatment success | 0
  Missing for partial treatment success | 0
  Complete response for treatment failure | 0
  Partial response for treatment failure | 0
  Stable disease for treatment failure | 8
  Progressive disease for treatment failure | 10
  Unknown for treatment failure | 1
  Missing for treatment failure | 20

5. Secondary Outcome: The Overall Safety and Tolerability of Pasireotide
Description: Safety assessments consisted of recording all AEs and serious adverse events (SAEs), the regular monitoring of hematology, blood chemistry, vital signs, physical condition and body weight.
Time Frame: At least 15 days
Population: The safety population consisted of all patients who received study drug (i.e. who started the pasireotide injections) and was thus identical to the Intent to treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Pasireotide (Any Dose)
Number analyzed (Participants) | 44
Participants
  Death | 1
  Serious or Significant Events | 23
  Serious Adverse Events (SAEs) | 14
  Discontinued due to Adverse Events (AEs) | 12

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: The safety population consisted of all patients who received study drug. Dosing began at 150μg twice daily (300μg daily) and went up to 1200μg twice daily (2400μg daily). Through the duration of the study the 45 patients started at 300μg-≤900μg /day, 43 patients proceeded to >900μg-≤1500μg/day and 31 patients proceeded to >1500μg -≤2400μg/day.
Groups:
- Pasireotide 300 ≤ 900 μg: Pasireotide 300 ≤ 900 μg / day
- Pasireotide > 900 ≤ 1500 μg: Pasireotide > 900 ≤ 1500 μg / day
- Pasireotide > 1500 ≤ 2400 μg: Pasireotide > 1500 ≤ 2400 μg / day
Arm/Group | Pasireotide 300 ≤ 900 μg | Pasireotide > 900 ≤ 1500 μg | Pasireotide > 1500 ≤ 2400 μg
Serious Adverse Events (participants affected / at risk) | 3/45 | 3/43 | 10/31
Other Adverse Events (participants affected / at risk) | 24/45 | 20/43 | 21/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide 300 ≤ 900 μg (N=45) | Pasireotide > 900 ≤ 1500 μg (N=43) | Pasireotide > 1500 ≤ 2400 μg (N=31)
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Hepatic artery embolism (Hepatobiliary disorders) | 0 | 0 | 2
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide 300 ≤ 900 μg (N=45) | Pasireotide > 900 ≤ 1500 μg (N=43) | Pasireotide > 1500 ≤ 2400 μg (N=31)
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 7 | 2
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 6
Flatulence (Gastrointestinal disorders) | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 7 | 8 | 2
Steatorrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2
Fatigue (General disorders) | 6 | 2 | 7
Oedema peripheral (General disorders) | 1 | 3 | 3
Cystitis (Infections and infestations) | 0 | 0 | 2
Weight decreased (Investigations) | 7 | 6 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 2

LIMITATIONS AND CAVEATS:
No formal statistical comparisons were performed for this study. Summary statistics were provided to compare the different doses administered for the primary and secondary endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.